CLINICAL TRIAL: NCT06935188
Title: Dalpicilib Plus Cetuximab Compared With Cetuximab Alone in Patients With HPV-negative, Anti-PD-1-resistant Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma: An Open Label, Randomized Controlled, Phase II Trial
Brief Title: Dalpicilib Plus Cetuximab Compared With Cetuximab Alone in HPV-negative, Anti-PD-1-resistant R/M HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, ren guoxin, Dr., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dawn-01 study
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dalpicilib combined with cetuximab (Experimental): The participants receive cetuximab in combination with Dalpiciclib until termination criteria are met. Participants receive cetuximab intravenously at a dose of 500 mg/m2 biweekly, or an initial dose of 400 mg/m² followed by weekly maintenance dose of 250 mg/m2. Dalpiciclib is administered orally at a dose of 150 mg once daily for 21 consecutive days, followed by a 7-day break. Each 28 days were deemed as a treatment cycle. If the patient vomits or misses a dose, it should not be made up on the same day. The next dose should be taken as usual.
  Interventions: Drug: Dalpicilib combined with cetuximab
- cetuximab (Active Comparator): The participants receive cetuximab alone until termination criteria are met. Participants receive cetuximab intravenously at a dose of 500 mg/m2 biweekly, or an initial dose of 400 mg/m² followed by weekly maintenance dose of 250 mg/m2.
  Interventions: Drug: cetuximab

INTERVENTIONS:
Drug: Dalpicilib combined with cetuximab — The participants receive cetuximab in combination with Dalpiciclib until termination criteria are met. Participants receive cetuximab intravenously at a dose of 500 mg/m2 biweekly, or an initial dose of 400 mg/m² followed by weekly maintenance dose of 250 mg/m2. Dalpiciclib is administered orally at a dose of 150 mg once daily for 21 consecutive days, followed by a 7-day break. Each 28 days were deemed as a treatment cycle. If the patient vomits or misses a dose, it should not be made up on the same day. The next dose should be taken as usual.
  Arms: Dalpicilib combined with cetuximab
Drug: cetuximab — The participants receive cetuximab alone until termination criteria are met. Participants receive cetuximab intravenously at a dose of 500 mg/m2 biweekly, or an initial dose of 400 mg/m² followed by weekly maintenance dose of 250 mg/m2.
  Arms: cetuximab

SUMMARY:
This study is a single center, randomized controlled, prospective phase II clinical trial to evaluate the efficacy and safety of cetuximab combined with dalpicilib compared to cetuximab monotherapy in patients with HPV-negative, anti-PD-1-resistant recurrent or metastatic head and neck squamous cell carcinoma. The participants would receive cetuximab combined with dalpicilib or cetuximab monotherapy until termination criteria are met.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, both sexes.
* Patients with histologically confirmed post-surgical recurrent/metastatic or locally advanced inoperable surgically resectable squamous cell carcinoma of the head and neck with measurable lesions (spiral CT scan ≥ 10 mm, meeting RECIST 1.1 criteria).
* Have received at least 1 cycle of prior PD-1 immunotherapy with imaging confirmation of progression or clinician determination of no continued benefit from treatment; provided that this is completed at least 4 weeks prior to the first dose of study drug and all associated toxic events have returned to normal or grade I or less as defined by CTCAE 4.03 classification.
* HPV viral testing determined to be negative, using the IHC method.
* Availability of tumor tissue (paraffin specimens less than 2 years old or fresh tumor tissue) for detection of PD-L1 and CDK4-related genes.
* ECOG score of 0 or 1.
* Expected survival of ≥ 12 weeks.
* Normal major organ function within 2 weeks prior to treatment, i.e., meeting the following criteria：Bone marrow function: hemoglobin ≥ 100 g/L without transfusion or colony-stimulating factor support therapy, white blood cell count ≥ 4.0*10^9/L or neutrophil count ≥ 2.0*10^9/L, and platelet count ≥ 100*10^9/L; Liver: serum total bilirubin level ≤ 1.5 times the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.5 times the upper limit of normal; Renal: blood creatinine level below 1.5 times the upper limit of normal or creatinine clearance ≥ 60 ml/min and urea nitrogen ≤ 200 mg/L; Urine protein <+, or if urine protein + then total 24-hour protein must be <500mg; Blood glucose: within normal range and/or with diabetes in treatment but under stable glycemic control; Pulmonary function: baseline FEV1 of at least 2L; if baseline FEV1 <2L then FEV1 >800ml expected post-surgery as assessed by a surgical specialist; Cardiac function: no myocardial infarction within 1 year; no unstable angina; no symptomatic severe arrhythmias; no cardiac insufficiency.

Exclusion Criteria:

* Patients previously treated with cetuximab or other anti-EGFR monoclonal antibodies or small molecule tyrosine kinase inhibitors.
* Patients who are currently receiving antineoplastic therapy.
* Patients who have participated or are participating in a clinical trial of another drug/therapy within 4 weeks prior to the first dose of the study drug.
* Patients who have received hematopoietic stimulating factors, such as granulocyte colony-stimulating factor (G-CSF), erythropoietin, etc., within 1 week prior to the first dose of the study drug.
* Positive HIV antibody or syphilis spirochete antibody test results.
* Patients with active hepatitis B or C: If positive for HBsAg or HBcAb, additional HBV DNA testing (results above the upper limit of the normal range). If HCV antibody test result is positive, add HCV RNA test (result above the upper limit of the normal range).
* Known hypersensitivity to recombinant humanized EGFR monoclonal antibody drugs and their components.
* Massive pleural or ascites fluid with clinical symptoms and requiring symptomatic management.
* Active lung disease (interstitial pneumonia, pneumonia, obstructive lung disease, asthma) or a history of active tuberculosis.
* Has any uncontrollable clinical problem, including but not limited to: Persistent or active (severe) infection; Poorly controlled diabetes mellitus; Cardiac disease (Class III/IV congestive heart failure or heart block as defined by the New York Heart Association); Deep vein thrombosis or pulmonary embolism; myocardial infarction; severe or unstable arrhythmia or angina; percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass grafting; cerebrovascular accident, transient ischemic attack, cerebral embolism within 6 months prior to first dose.
* Previous stem cell transplantation or organ transplantation.
* Those with a history of psychotropic substance abuse and unable to abstain or a history of psychiatric disorders.
* Other serious, acute or chronic medical conditions or abnormalities in laboratory tests that, in the judgment of the investigator, may increase the risk associated with study participation or may interfere with the interpretation of study results.
* Patients who, in the judgment of the investigator, have poor compliance or other conditions that make them unsuitable for participation in this trial.
* Patients with a history of other malignancies within five years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival Per RECIST 1.1 | 12 months
  PFS was defined as the time from enrollment to the first documented PD per RECIST 1.1, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD

SECONDARY OUTCOMES:
objective response rate | 12 months
  ORR was defined as the percentage of participants in the analysis population who have a Complete Response (CR:
  disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1.
overall survival | 12 months
  OS was defined as the time from enrollment to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up.
Number of Participants Experiencing an Adverse Event (AE) | 12 months
  An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants that experienced at least one AE was reported for each treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Yue He, Principal Investigator — the Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- the Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China